CLINICAL TRIAL: NCT00678704
Title: A Randomized, Placebo-controlled, Double-blind, Multi-centre, Parallel Group Study to Investigate the Efficacy and Safety of BAY 38-9456 in Males With Diabetes Suffering From Erectile Dysfunction
Brief Title: BAY38-9456 - Pivotal Trial for Diabetes Patient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100607
Record Dates: First submitted 2008-04-01; First posted 2008-05-15 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction; Diabetes Mellitus
Keywords: Vardenafil; PDE5 inhibitor; Erectile Dysfunction; Diabetes Mellitus; Sexual Dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus; Sexual Dysfunction, Physiological | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — BAY 38-9456 10 mg tablet prior to intercourse on demand
  Arms: Arm 1
Drug: Levitra (Vardenafil, BAY38-9456) — BAY 38-9456 20 mg tablet prior to intercourse on demand
  Arms: Arm 2
Drug: Placebo — Placebo tablet prior to intercourse on demand
  Arms: Arm 3

SUMMARY:
The superiority of BAY 38-9456 10 mg and 20 mg regimens to placebo, and of 20 mg to 10 mg was confirmed in patients with diabetes mellitus suffering from erectile dysfunction. There was no large difference in incidence rate of drug-related adverse events between 10 mg and 20 mg regimens. Overall the tolerability was considered good with both regimens.

ELIGIBILITY:
Inclusion Criteria:

* Male with erectile dysfunction for more than 3 years according to the National Institutes of Health (NIH) Consensus Statement (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance)
* Diabetes for more than 3 years

Exclusion Criteria:

* Following to the labeling of Japanese package insert for vardenafil 5/10 mg, except for the highest dose
* Spinal cord injury
* History of surgical prostatectomy (excluding TURP)
* Patients with an HbA1c > 12% at Visit 1
* Use of nitrates
* Use of potent CYP3a4 inhibitors
* Severe liver disease
* Presence of Peyronie's Disease

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 790 (Actual)
Dates: Start 2004-01; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The Erectile Function (EF) domain score of IIEF calculated as the sum of scores from Questions 1 to 5 and 15 | At 12 weeks after start of study drug administration using data at LOCF to account for dropouts

SECONDARY OUTCOMES:
The Global Assessment Question | At 4, 8, 12 weeks after start of study drug administration and LOCF
The IIEF EF domain score | At 4, 8, 12 weeks after start of study drug administration
IIEF domain scores other than the EF domain score[intercourse satisfaction (Q6 to Q8), overall satisfaction (Q13, Q14), orgasmic function (Q9, Q10), sexual desire (Q11, Q12)] | At 4, 8, 12 weeks after start of study drug administration and LOCF
Scores of Questions 1 to 15 on the IIEF Questionnaire | At 4, 8, 12 weeks after start of study drug administration and LOCF
Patient's diary response concerning hardness of erection, maintenance of erection, satisfaction with overall hardness of erection, ability of insertion, overall satisfaction with sexual experience and ejaculation | At 4, 8, 12 weeks after start of study drug administration and LOCF
Safety data | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer